CLINICAL TRIAL: NCT06086444
Title: The Effectiveness of Tranexamic Acid in Abdominoplasty Plastic Surgery.
Brief Title: Tranexamic Acid in Abdominoplasty.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16/2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-01

CONDITIONS: Abdominal Wall Defect; Hemorrhage; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Sodium Chloride; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline for intravenous administration.
  Interventions: Drug: Placebo
- Tranexamic acid (Active Comparator): Tranexamic Acid for intravenous administration.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Placebo — 100 mL of normal saline. Administered intravenously at least 10 minutes prior to skin incision.
  Other Names: 0.9% sodium chloride
  Arms: Placebo
Drug: Tranexamic acid — Tranexamic Acid (10mg/kg), diluted in 100 ccs of normal saline. Administered intravenously at least 10 minutes before skin incision.
  Other Names: TXA
  Arms: Tranexamic acid

SUMMARY:
The investigators prepared a novel tranexamic acid (TXA) study designed to estimate the quantity of blood loss in patients undergoing abdominoplasty surgery. This study aims to quantify blood loss during abdominoplasty with and without TXA. The central hypothesis is that TXA administration reduces blood loss and fibrinolysis in patients undergoing abdominoplasty surgery.

DETAILED DESCRIPTION:
Tranexamic acid (TXA) treatment is increasingly emphasized in plastic surgery because TXA inhibits fibrinolysis. Increased clot stability offers the possibility of preventing blood loss (prevention) and mitigating ongoing hemorrhage. TXA therapy has been principally studied in populations; the results of studies in plastic surgery still need to be improved.

Tranexamic acid is an antifibrinolytic agent that acts as a competitive inhibitor at the lysine binding sites of plasminogen and inhibits the ability of protease plasmin to cleave the fibrin clot. In large randomized controlled trials, it has been reported to be effective in decreasing perioperative blood loss in various circumstances, primarily involving trauma patients.

The investigators designed a randomized placebo-controlled trial comparing TXA dosing before incision for abdominoplasty. The purpose is to quantify blood loss during plastic surgery with and without TXA.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled abdominoplasty
* ASA 1 or 2
* age >18 and <75 years

Exclusion Criteria:

* BMI <20 or >35 kg/m2
* ASA 3 or > 3
* medical history of thromboembolism
* history of hematological disease
* treatment with aspirin 14 days before the procedure
* treatment with anticoagulants 5 days before the procedure
* epilepsy
* allergy to tranexamic acid
* coagulation disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Blood loss volume | 24 hours after surgery
  Total blood volume loss will be calculated in milliliters.

SECONDARY OUTCOMES:
HBG | 24 hours after surgery
  Hemoglobin level measured before and 24 hours after surgery
D-dimer | 24 hours after surgery
  D-dimer level measured before and 24 hours after surgery
Fibrinogen | 24 hours after surgery
  Fibrinogen level measured before and 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, Ph.D., Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

REFERENCES:
- [Derived] Kolasinski J, Reysner T, Kolenda M, Kolacz S, Reysner M. Efficacy and safety of intravenous tranexamic acid in elective abdominoplasty: A randomized, triple-blinded, placebo-controlled clinical trial. J Plast Reconstr Aesthet Surg. 2025 Dec 5;113:693-699. doi: 10.1016/j.bjps.2025.11.055. Online ahead of print. PMID 41520615